CLINICAL TRIAL: NCT04526626
Title: Endovenous Radiofrequency Ablation Versus High Ligation and Striping for Treatment of Varicose Veins: a Prospective Controlled Trial
Brief Title: Endovenous RFA Versus Ligation and Striping for Varicose Veins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKUSZH201901013
Record Dates: First submitted 2020-03-25; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Radiofrequency ablation; High ligation and striping
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- High ligation and stripping (Experimental): High ligation and stripping of long saphenous vein is the traditional standard procedure for the treatment of varicose veins
  Interventions: Device: Radiofrequency ablation for treatment of lower limb varicose veins (ClosureFast, Medtronic)

INTERVENTIONS:
Device: Radiofrequency ablation for treatment of lower limb varicose veins (ClosureFast, Medtronic) — Thermal injury to long saphenous vein
  Other Names: ClosureFast, Medtronic

SUMMARY:
Varicose vein is a common chronic disease affecting patient's quality of life. High ligation and stripping of the long saphenous vein is the traditional operation for varicose vein. The radiofrequency ablation (RFA) device used for treatment of varicose vein has been available in China since 2014. There are few studies comparing RFA and stripping in the treatment of varicose vein. This study was to investigate the outcomes of RFA and stripping for varicose vein. Patients with varicose veins will be prospectively allocated to RFA group and stripping group. Ultrasound follow-up will be performed to assess recanalization of long saphenous vein at 1 month, 3, 6 and 12 months. Recurrence of varicose vein and improvement of symptoms will also be evaluated. The primary endpoints are technical success, complications and recurrence of varicose vein. Secondary endpoints are duration of operation, blood loss, recovery time, venous clinical severity score, and medical cost. The treatment outcomes will be compared between the RFA group and stripping group. RFA is comparable to traditional stripping in the treatment of varicose vein, however, it is associated quick recovery, lower incidence of complications and higher medical cost.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of long saphenous varicose veins

Exclusion Criteria:

* Contraindicated to operation due to severe comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | up to 24 months
  Occlusion of the long saphenous vein
Complications | 2 weeks after operation
  Deep vein thrombosis, skin burn
Recurrence of varicose vein | up to 24 months
  Recurrence of varicose vein

CONTACTS AND LOCATIONS:
Overall Officials: Hailei Li, M.D, Ph.D, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- University of Hong Kong Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No